CLINICAL TRIAL: NCT01048853
Title: Conservative Surgery for Women With Low-Risk, Early Stage Cervical Cancer
Brief Title: Conservative Surgery in Treating Patients With Low-Risk Stage IA2 or IB1 Cervical Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: < 75% participation
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0118; NCI-2012-01254 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2008-0118 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2010-01-12; First posted 2010-01-14 (Estimated); Results first posted 2025-11-26 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Cervical Adenocarcinoma; Cervical Squamous Cell Carcinoma, Not Otherwise Specified; Stage IA2 Cervical Cancer AJCC v6 and v7; Stage IB1 Cervical Cancer AJCC v6 and v7
MeSH Terms: interventions — Salpingo-oophorectomy; Sentinel Lymph Node Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (conservative surgery) (Experimental): Patients undergo a complete lymphatic mapping with sentinel lymph node biopsy and/or pelvic lymph node dissection. If future fertility is no longer desired, patients also undergo hysterectomy with or without bilateral salpingo-oophorectomy.
  Interventions: Procedure: Lymph Node Mapping; Other: Quality-of-Life Assessment; Procedure: Salpingo-Oophorectomy; Procedure: Sentinel Lymph Node Biopsy; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Procedure: Lymph Node Mapping — Undergo lymphatic mapping with sentinel lymph node biopsy
  Other Names: lymphatic mapping
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Procedure: Salpingo-Oophorectomy — Undergo hysterectomy with or without salpingo-oophorectomy
Procedure: Sentinel Lymph Node Biopsy — Undergo lymphatic mapping with sentinel lymph node biopsy
  Other Names: Sentinel Node Biopsy; Sentinel node biopsy alone; SLNB; SNB
Procedure: Therapeutic Conventional Surgery — Undergo hysterectomy with or without salpingo-oophorectomy

SUMMARY:
This clinical trial studies conservative surgery in treating patients with low-risk stage IA2 or IB1 cervical cancer. Conservative surgery is a less invasive type of surgery for early stage cervical cancer and may have fewer side effects and improve recovery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety and feasibility of performing conservative surgery in women with stage IA2 or IB1 carcinoma of the cervix with favorable pathologic features.

SECONDARY OBJECTIVES:

I. To estimate the cervix cancer recurrence rate at 2 years in women treated with conservative surgery for stage IA2 or IB1 carcinoma of the cervix with favorable pathologic features.

II. To compare pelvic lymph node involvement in patients undergoing conservative surgery with historical data from matched patients treated with radical hysterectomy.

III. To estimate the sensitivity of sentinel lymph node biopsy in the determination of pelvic lymph node metastases in this group of patients.

IV. To compare the treatment-associated morbidity in patients undergoing conservative surgery with historical data from matched patients treated with radical hysterectomy.

V. To assess quality of life factors, sexual functioning, symptoms and satisfaction with healthcare decisions in this group of patients.

OUTLINE:

Patients undergo a complete lymphatic mapping with sentinel lymph node biopsy and/or pelvic lymph node dissection. If future fertility is no longer desired, patients also undergo hysterectomy with or without bilateral salpingo-oophorectomy.

After completion of study treatment, patients are followed up every 3 months for 2 years and then yearly for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma of the cervix (any grade) or histologically confirmed grade 1 or 2 adenocarcinoma of cervix
* International Federation of Gynecology and Obstetrics (FIGO) stage IA2 or IB1 disease
* Tumor diameter =< 2 cm on physical exam and on imaging studies
* No lymphovascular space invasion (LVSI) present on biopsy or previous cone
* Less than 10 mm of cervical stromal invasion
* Cone margins and endocervical curettage (ECC) specimen negative for invasive cancer, cervical intraepithelial neoplasia (CIN) II, CIN III or adenocarcinoma-in-situ; (a negative margin is defined as no invasive cancer within 1.0 mm of both the endocervical and ectocervical margins and no adenocarcinoma in situ [AIS] or CIN II or CIN III at the inked or cauterized margin; one repeat cone and ECC permitted)
* Patients are eligible for the study when a cone and ECC are performed prior to pre-enrollment in the study, and pathologic eligibility criteria are met; the cone and ECC must be performed within 12 weeks prior to pre-enrollment in the study; if the cone and ECC performed prior to pre-enrollment do not meet the pathologic criteria, patients may be pre-enrolled and are allowed 1 repeat cone & ECC after pre-enrollment in order to meet pathologic eligibility criteria
* Patients must sign an approved informed consent document
* If patient is of childbearing potential, she must have a negative blood or urine pregnancy test within 14 days of surgical treatment on study
* Imaging with positron emission tomography (PET) scan, computed tomography (CT) scan of the abdomen and pelvis, and/or magnetic resonance imaging (MRI) of the abdomen and pelvis must be performed and negative for metastatic disease within 12 weeks of enrollment

Exclusion Criteria:

* Clear cell, neuroendocrine, adenosquamous, serous carcinoma or other high-risk histologies
* Grade 3 adenocarcinoma
* FIGO stage IA1, IB2, II, III or IV disease
* Tumors > 2 cm in diameter on physical exam or imaging studies
* Presence of LVSI
* Greater than or equal to 10 mm of cervical stromal invasion
* Cone margins or ECC specimen positive for invasive cancer, CIN II, CIN III or adenocarcinoma-in-situ (one repeat cone permitted)
* Neoadjuvant radiation therapy or chemotherapy for cervical cancer
* Patients unwilling or unable to provide informed consent for the study
* Evidence of metastatic disease on PET, CT, and/or MRI performed within 12 weeks of enrollment
* Patients who have had a simple hysterectomy (cut through hysterectomy)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2010-04-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Schmeler, Principal Investigator — M.D. Anderson Cancer Center
Locations (20):
- United States (11):
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Northwell Health Imbert Cancer Center, Bay Shore, New York
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - The Woman's Hospital of Texas, Houston, Texas
  - MD Anderson in Katy, Houston, Texas
  - MD Anderson League City, Nassau Bay, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - MD Anderson in The Woodlands, The Woodlands, Texas
- Argentina (3):
  - Hospital Italiano of Buenos Aires, Buenos Aires
  - Hospital Israelita Buenos Aires, Buenos Aires
  - Instituto de Oncologia Angel H Roffo, Buenos Aires
- Royal Women's Hosptial, Melbourne, Victoria, Australia
- Hosptial de Cancer de Barretos, Barretos, São Paulo, Brazil
- Instituto Nacional De Cancerologia, Bogotá, Colombia
- Instituto Nacional De Cancerologia de Mexico, Mexico City, Tlalpan, Mexico
- Instituto Nacional de Enfermedades Neoplasicas, Lima, Peru
- King Chulalongkorn University, Bangkok, Pathumwan, Thailand

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Fertility Sparing: Conization followed by lymph node assessment only
- Conization + Hysterectomy + Lymph Node Assessment: Conization followed by hysterectomy and lymph node assessment
- Simple Hysterectomy: Inadvertent simple hysterectomy followed by lymph node dissection
Period: Overall Study
Arm/Group | Fertility Sparing | Conization + Hysterectomy + Lymph Node Assessment | Simple Hysterectomy
Started | 44 | 40 | 16
Completed | 42 | 36 | 16
Not Completed | 2 | 4 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fertility Sparing | Conization + Hysterectomy + Lymph Node Assessment | Simple Hysterectomy | Total
Number analyzed (Participants) | 44 | 40 | 16 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 44 | 39 | 16 | 99
  >=65 years | 0 | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 31 [22 to 44] | 43 [24 to 66] | 47 [31 to 64] | 39 [22 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 40 | 16 | 100
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 22 | 5 | 52
  Not Hispanic or Latino | 14 | 11 | 7 | 32
  Unknown or Not Reported | 5 | 7 | 4 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 2 | 3
  White | 28 | 25 | 12 | 65
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 13 | 13 | 2 | 28
Region of Enrollment [Number; unit: participants]
  Colombia | 4 | 8 | 2 | 14
  Argentina | 6 | 1 | 0 | 7
  United States | 17 | 13 | 10 | 40
  Brazil | 10 | 6 | 3 | 19
  Mexico | 1 | 3 | 0 | 4
  Thailand | 1 | 0 | 0 | 1
  Australia | 0 | 1 | 0 | 1
  Peru | 4 | 8 | 1 | 13
  Italy | 1 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety and Feasibility of Performing Conservative Surgery in Women With Stage IA2 or IB1 Carcinoma of the Cervix With Favorable Pathologic Features
Description: The proposed treatment strategy will be considered not feasible if the immediate failure rate is more than 3%. The immediate failure rate, defined as residual disease in the simple hysterectomy specimen of women who underwent conization followed by simple hysterectomy and lymph node assessment.
Time Frame: Approximately 9 years
Population: Fertility Sparing - hysterectomy not performed. Simple Hysterectomy - hysterectomy performed prior to study enrollment.
  Conization + hysterectomy + lymph node assessment group was only group assessed as Fertility Sparing did not have hysterectomy and the Simple Hysterectomy group had hysterectomy performed prior to study enrollment making them inevaluable.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Fertility Sparing | Conization + Hysterectomy + Lymph Node Assessment | Simple Hysterectomy
Number analyzed (Participants) | 0 | 40 | 0
percentage of participants |  | 2.5 [0.2 to 7.2] |

2. Secondary Outcome: Cervix Cancer Recurrence Rate at 2 Years in Women Treated With Conservative Surgery for Stage IA2 or IB1 Carcinoma of the Cervix With Favorable Pathologic Features
Description: Recurrence rate was estimated and was measured from the date of surgery to the earliest date of the last clinic visit, date of first recurrence, or date of death.
Time Frame: 2 years
Population: Only 42 participants out of 44 in the fertility sparing group were evaluated; 1 participant expired following the surgical procedure and 1 participant was lost to follow up prior to the 2 year interval. In the conization + hysterectomy group, 4 participants of the 40 in this group were lost to follow up prior to the 2 year interval.
Measure: Number; unit: percentage of participants
Arm/Group | Fertility Sparing | Conization + Hysterectomy + Lymph Node Assessment | Simple Hysterectomy
Number analyzed (Participants) | 42 | 36 | 16
percentage of participants | 2.4 | 0 | 12.5

3. Secondary Outcome: Number of Participants With All-Cause Mortality
Description: Total patient morbidity within 30 days following conservative surgery
Time Frame: Approximately 9 years
Measure: Count of Participants; unit: Participants
Arm/Group | Fertility Sparing | Conization + Hysterectomy + Lymph Node Assessment | Simple Hysterectomy
Number analyzed (Participants) | 44 | 40 | 16
Participants | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were reported for approximately 9 years
Arm/Group | Fertility Sparing | Conization + Hysterectomy + Lymph Node Assessment | Simple Hysterectomy
All-Cause Mortality (participants affected / at risk) | 1/44 | 0/40 | 0/16
Serious Adverse Events (participants affected / at risk) | 5/44 | 3/40 | 1/16
Other Adverse Events (participants affected / at risk) | 5/44 | 5/40 | 4/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fertility Sparing (N=44) | Conization + Hysterectomy + Lymph Node Assessment (N=40) | Simple Hysterectomy (N=16)
Thrombolic event (General disorders) | 1 | 0 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Uterine obstruction (Renal and urinary disorders) | 2 | 0 | 0
Numbness right leg (Nervous system disorders) | 1 | 0 | 0
Wound dehiscence (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Pelvic infection (Reproductive system and breast disorders) | 0 | 1 | 0
Brusing/swelling in mons (Reproductive system and breast disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fertility Sparing (N=44) | Conization + Hysterectomy + Lymph Node Assessment (N=40) | Simple Hysterectomy (N=16)
Bladder anastomotic leak (Renal and urinary disorders) | 0 | 1 | 0
Abdominal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Uterine hemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Pelvic pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Hematoma (General disorders) | 0 | 1 | 0
Edema limbs (General disorders) | 1 | 0 | 0
Lymphedema (General disorders) | 0 | 0 | 1
Abnormal area of vagina noted (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1
Vascular injury (Vascular disorders) | 1 | 0 | 0
Left groin swelling (General disorders) | 0 | 1 | 0
Wound complication (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-29): https://cdn.clinicaltrials.gov/large-docs/53/NCT01048853/Prot_SAP_000.pdf
  • Informed Consent Form (2020-02-05): https://cdn.clinicaltrials.gov/large-docs/53/NCT01048853/ICF_001.pdf